CLINICAL TRIAL: NCT04315948
Title: Multi-centre, Adaptive, Randomized Trial of the Safety and Efficacy of Treatments of COVID-19 in Hospitalized Adults
Brief Title: Trial of Treatments for COVID-19 in Hospitalized Adults
Acronym: DisCoVeRy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C20-15; 101015736 (Other Grant/Funding Number: H2020-EU.3.1.3.)
Record Dates: First submitted 2020-03-13; First posted 2020-03-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Corona Virus Infection
Keywords: COVID-19; SARS-CoV-2; Pneumonia
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Pneumonia | interventions — remdesivir; Lopinavir; Interferon beta-1a; Hydroxychloroquine; Standard of Care; cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Intervention Model Description: From March 22, 2020 to May 24, 2020, the study randomized participants 1:1:1:1:1 to standard of care alone (control) or with investigational product added.
  From May 24, 2020 to June 29, 2020, the study randomized participants 1:1:1:1 to standard of care alone (control) or with investigational product added.
  From June 29, 2020 to January 19,2021, the study randomized participants 1:1 to standard of care alone (control) or with investigational product added.
  Since April, 2021, the study will randomize participants 1:1 to standard of care with placebo (control) or standard of care with investigational product added.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * the treatment arm SOC + hydroxychloroquine has been ceased since May 24, 2020;
  * the treatment arm SOC + lopinavir / Ritonavir and lopinavir / ritonavir + interferon ß-1a has been ceased since June 29, 2020
  * the treatment arm SOC + remdesivir has been ceased since January 19, 2021
  * the treatment arm SOC + AZD7442
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Remdesivir (Experimental): Remdesivir will be administered as a 200 mg intravenous loading dose on Day 1, followed by a 100 mg once-daily intravenous maintenance dose for the duration of the hospitalization up to a 10 days total course.
  n=475
  Interventions: Drug: Remdesivir; Other: Standard of care
- Lopinavir/ritonavir (stopped on June 29, 2020) (Experimental): Lopinavir/ritonavir (400 lopinavir mg/100 mg ritonavir) will be administered every 12 h for 14 days in tablet form. For patients who are unable to take medications by mouth, the lopinavir/ritonavir (400 lopinavir mg/100 mg ritonavir) will be administered as a 5-ml suspension every 12 h for 14 days via a pre-existing or newly placed nasogastric tube.
  n=620
  Interventions: Drug: Lopinavir/ritonavir; Other: Standard of care
- Lopinavir/ritonavir plus Interferon ß-1a (stopped on June 29) (Experimental): Lopinavir/ritonavir (400 lopinavir mg/100 mg ritonavir) will be administered every 12 h for 14 days in tablet form. For patients who are unable to take medications by mouth, the lopinavir/ritonavir (400 lopinavir mg/100 mg ritonavir) will be administered as a 5-ml suspension every 12 h for 14 days via a pre-existing or newly placed nasogastric tube.
  Interferon ß1a will be administered subcutaneously at the dose of 44 µg for a total of 3 doses in 6 days (day 1, day 3, day 6).
  n=620
  Interventions: Drug: Lopinavir/ritonavir; Drug: Interferon Beta-1A; Other: Standard of care
- Hydroxychloroquine (stopped on May 24, 2020) (Experimental): Hydroxychloroquine will be administered orally as a loading dose of 400 mg twice daily for one day followed by 400 mg once daily for 9 days. The loading dose of hydroxychloroquine through a nasogastric tube will be increased to 600 mg twice a day for one day, followed by a maintenance dose of 400 mg once a day for 9 days n=620
  Interventions: Drug: Hydroxychloroquine; Other: Standard of care
- Standard of care alone (Active Comparator): Standard of care alone before March, 2021.
  Interventions: Other: Standard of care
- AZD7442 (Experimental): Participants randomized to the AZD7442 group will receive a total dose of 600 mg AZD7442 via a co-administered (300 mg AZD8895 and 300 mg AZD1061) single IV infusion on Day 1.
  n=620
  Interventions: Other: Standard of care; Drug: AZD7442
- Standard of care with placebo (Active Comparator): Standard of care with placebo since April, 2021 n=620
  Interventions: Other: Standard of care; Other: Placebo

INTERVENTIONS:
Drug: Remdesivir — The lyophilized formulation of Remdesivir is a preservative-free, white to off-white or yellow, lyophilized solid containing 100 mg of Remdesivir to be reconstituted with 19 mL of sterile water for injection and diluted into IV infusion fluids prior to IV infusion. Following reconstitution, each vial contains a 5 mg/mL Remdesivir concentrated solution with sufficient volume to allow withdrawal of 20 mL (100 mg of remdesivir). It is supplied as a sterile product in a single-use, 30 mL, Type 1 clear glass vial.
  Arms: Remdesivir
Drug: Lopinavir/ritonavir — The oral tablets of lopinavir/ritonavir contain 200 mg lopinavir, 50 mg ritonavir. They have a yellow colour, film-coated, ovaloid shape debossed with the "a" logo and the code KA. The oral solution for patients who cannot swallow is a light yellow to orange colored liquid containing 400 mg lopinavir and 100 mg ritonavir per 5 mL (80 mg lopinavir and 20 mg ritonavir per mL).
  Arms: Lopinavir/ritonavir (stopped on June 29, 2020); Lopinavir/ritonavir plus Interferon ß-1a (stopped on June 29)
Drug: Interferon Beta-1A — IFN-ß-1a is supplied as a sterile solution containing no preservative available in a prefilled syringe. It will be provided as a single-dose prefilled graduated syringe with 44 µg per 0.5 mL. The liquid should be clear to slightly yellow. Do not use if the liquid is cloudy, discolored or contains particles. Use a different syringe.
  Arms: Lopinavir/ritonavir plus Interferon ß-1a (stopped on June 29)
Drug: Hydroxychloroquine — Hydroxychloroquine is supplied as film-coated 200 mg tablets. Hydroxychloroquine sulfate tablets are presented as white or whitish, peanut-shaped, oblong or round film-coated tablets containing 200 mg of hydroxychloroquine sulfate (equivalent to 155 mg base).
  Arms: Hydroxychloroquine (stopped on May 24, 2020)
Other: Standard of care — Standard of care
Drug: AZD7442 — AZD7442 will be supplied as separate vials of AZD8895 and AZD1061 containing 150 mg colorless to slightly yellow, clear to opalescent solutions for injection.
  Arms: AZD7442
Other: Placebo — Since April, 2021, the placebo will be a 0.9% (w/v) NaCl solution for infusion also called saline. The placebo will be supplied as a single 10-mL, clear and colorless vial.
  Arms: Standard of care with placebo

SUMMARY:
DisCoVeRy is a randomized controlled trial among adults (≥18-year-old) hospitalized for COVID-19. This study is an adaptive, randomized, open or blinded, depending on the drug to be evaluated, clinical trial to evaluate the safety and efficacy of possible therapeutic agents in hospitalized adult patients diagnosed with COVID-19. The study is a multi-centre/country trial that will be conducted in various sites in Europe with Inserm as sponsor. The study will compare different investigational therapeutic agents to a control group managed with the SoC including corticosteroids and anticoagulants. There will be interim monitoring to allow early stopping for safety and to introduce new therapies as they become available. If one therapy proves to be superior to others in the trial, this treatment may become part of the SoC for comparison(s) with new experimental treatment(s).

In previous versions of the DisCoVeRy protocol, remdesivir, lopinavir/ritonavir with or without interferon ß-1a and hydroxychloroquine were evaluated as potential treatments for COVID-19. These treatments have been discontinued based on analyses review by both DSMC/DSMB, the Solidarity Executive Group and the DisCoVeRy steering committee.

This version of the protocol, therefore, describes a randomized blinded placebo-controlled trial among adults (≥18-year-old) hospitalized for COVID-19 that randomly allocates them (1:1 ratio) between 2 arms: SoC + placebo versus SoC + AZD7442.

Randomization will be stratified by region (according to the administrative definition in each country), antigenic status (positive or negative) obtained from the result of a rapid antigen test on nasopharyngeal swab performed at enrolment and vaccination initiation (yes or no).

The primary analyses will be conducted on patients with antigen-positive results. A positive antigenic test is evidence of high viral shedding consistent with a recently started or uncontrolled infection. Overall, the number of antigen-negative patients will be at most 30% of all included subjects. The number of patients with vaccination (partly or fully) will be limited to 20% of all participants, split evenly between antigen positive and antigen negative patients (i.e. vaccinated patients can make up at most 20% of antigene positive patients and 20% of antigene negative patients). Sensitivity analyses will be performed in all patients, stratified by antigenic status and vaccination initiation.

A global independent data and safety monitoring board (DSMB) monitors interim data to make recommendations about early study closure or changes to conduct, including adding or removing treatment arms. However, the current version of the protocol does not allow for efficacy or futility analysis, and the ability to add trial arms will be limited by the study being blinded and placebo-controlled during the investigation of AZD7442.

DETAILED DESCRIPTION:
DisCoVeRy is a randomized controlled trial among adults (≥18-year-old) hospitalized for COVID-19. This study is an adaptive, randomized, open or blinded, depending on the drug to be evaluated, clinical trial to evaluate the safety and efficacy of possible therapeutic agents in hospitalized adult patients diagnosed with COVID-19. The study is a multi-centre/country trial that will be conducted in various sites in Europe with Inserm as sponsor. The study will compare different investigational therapeutic agents to a control group managed with the SoC including corticosteroids and anticoagulants. There will be interim monitoring to allow early stopping for safety and to introduce new therapies as they become available. If one therapy proves to be superior to others in the trial, this treatment may become part of the SoC for comparison(s) with new experimental treatment(s).

In previous versions of the DisCoVeRy protocol, remdesivir, lopinavir/ritonavir with or without interferon ß-1a and hydroxychloroquine were evaluated as potential treatments for COVID-19. These treatments have been discontinued based on analyses review by both DSMC/DSMB, the Solidarity Executive Group and the DisCoVeRy steering committee.

This version of the protocol, therefore, describes a randomized blinded placebo-controlled trial among adults (≥18-year-old) hospitalized for COVID-19 that randomly allocates them (1:1 ratio) between 2 arms: SoC + placebo versus SoC + AZD7442.

Randomization will be stratified by region (according to the administrative definition in each country), antigenic status (positive or negative) obtained from the result of a rapid antigen test on nasopharyngeal swab performed at enrolment and vaccination initiation (yes if at least one injection of any vaccine against SARS-CoV-2 was reveived prior to enrolment whatever the delay or no).

The primary analyses will be conducted on patients with antigen-positive results. A positive antigenic test is evidence of high viral shedding consistent with a recently started or uncontrolled infection. Overall, the number of antigen-negative patients will be at most 30% of all included subjects. The number of patients with vaccination (partly or fully) will be limited to 20% of all participants, split evenly between antigen positive and antigen negative patients (i.e. vaccinated patients can make up at most 20% of antigene positive patients and 20% of antigene negative patients). Sensitivity analyses will be performed in all patients, stratified by antigenic status and vaccination initiation.

A global independent data and safety monitoring board (DSMB) monitors interim data to make recommendations about early study closure or changes to conduct, including adding or removing treatment arms. However, the current version of the protocol does not allow for efficacy or futility analysis, and the ability to add trial arms will be limited by the study being blinded and placebo-controlled during the investigation of AZD7442.

All subjects will undergo a series of efficacy and safety assessments, including laboratory assays.

Subjects will be assessed at baseline, and at Days 3, 8 and 15 while hospitalized. Patients will be contacted by phone at Day 15 for evaluation of the Primary Endpoint if they have been discharged prior to Day 15-, and 14-days following hospital discharge for efficacy assessment.

Further follow-up assessments will be organized at Days 29, 90, 180, 365 and 456.

If discharged from the hospital, days 29 and 90 assessments will be organized as outpatients' consultations for all. For Days 180 and 365 assessments, a subset of 25% of patients enrolled in centers with available resources and selected at Day 90 will be evaluated during a medical consultation, while the other will be contacted by phone. For Day 456, all patients will be contacted by phone.

Nasopharyngeal swabs (NP) or lower respiratory tract samples will be obtained at baseline (Day 1 pre-treatment) and at Days 3, 8, 15 (while hospitalized) and 29 (while hospitalized or, if discharged from the hospital, in the outpatient setting).

Blood samples will be obtained at baseline (Day 1 pre-treatment) and at Days 3, 8, 15 (while hospitalized), at Days 29 and 90, and at Days 180 and 365 (for the subset of patients evaluated during a medical consultation at these times).

Thoracic computed tomography (CT)-scan will be obtained at baseline, depending on the centre's imagery capacities.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥18 years of age at the time of enrolment
2. Hospitalized patients with any of the following criteria:

   1. the presence of pulmonary rales/crackles on clinical exam OR
   2. SpO2 ≤ 94% on room air OR
   3. requirement of supplementary oxygen including high flow oxygen devices or non-invasive ventilation
3. A time between onset of symptoms and randomization of less than 11 days
4. A positive SARS-CoV-2 PCR performed on a NP swab within the 5 days preceding randomization
5. The result of a rapid antigen test performed on a NP swab within the 6 hours preceding randomization
6. Contraceptive use by men or women.

   1. Male participants: Contraception for male participants is required; to avoid the transfer of any fluids, all male participants must use a condom from Day 1 and agree to continue for 90 days following administration of IMP.
   2. Female participants: Women of child-bearing potential must agree to use contraception for 365 days following administration of IMP

Exclusion Criteria:

1. Refusal to participate expressed by patient or legally authorized representative
2. Need for invasive mechanical ventilation and/or ECMO at the time of enrolment
3. Spontaneous blood ALT/AST levels > 5 times the upper limit of normal
4. Glomerular filtration rate (GFR) < 15 mL/min or requiring maintenance dialysis
5. Pregnancy or breast-feeding
6. Anticipated transfer to another hospital, which is not a study site within 72 hours following randomization
7. Known history of allergy or reaction to any component of the study drug formulation.
8. Previous hypersensitivity, infusion-related reaction, or severe adverse reaction following administration of monoclonal or polyclonal antibodies.
9. Any prior receipt of investigational or licensed other mAb/biologic indicated for the prevention of SARS-CoV-2 infection or COVID-19, and for those not vaccinated, expected receipt of vaccine in the 30 days following hospital discharge, according to current recommendation in each country.
10. Any medical condition which, in the judgment of the investigator, could interfere with the interpretation of the trial results or that preludes to protocol adherence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1552 (Actual)
Dates: Start 2020-03-22 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects reporting each severity rating on a 7-point ordinal scale | Day 15
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities;
  3. Hospitalized, not requiring supplemental oxygen;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  6. Hospitalized, on invasive mechanical ventilation or ECMO;
  7. Death.

SECONDARY OUTCOMES:
Status on an ordinal scale | Days 29, 90, 180 and 365
  Percentage of subjects reporting each severity rating on a 7-point on an ordinal scale
National Early Warning Score 2 (NEWS-2 score) | Days 3, 8, 15, and 29
  Change from baseline in NEWS-2.
Number of oxygenation free days in the first 28 days | 29 days
Incidence of new oxygen use, non-invasive ventilation or high flow oxygen devices during the trial. | 29 days
Ventilator free days in the first 28 days | 29 days
Incidence of new mechanical ventilation use during the trial. | 29 days
Need for mechanical ventilation or death by Day 15 | Day 15
  Proportion of patients with mechanical ventilation or death at day 15
Hospitalization | 29 days
  Time to hospital discharge (days).
Mortality | In hospital, Days 29, 90, 180, 365, 456
  Rate of mortality
Occurrence of new hospitalization | Days 90, 180 and 365
Occurrence of confirmed re-infection with SARS-CoV-2 | Days 90, 180 and 365
Cumulative incidence of serious adverse events (SAEs) | 29 days
Cumulative incidence of Grade 1- 2 hypersensitivity- related and infusion related AEs until D29 visit | 29 days
Cumulative incidence of Grade 3 and 4 adverse events (AEs) | 29 days
Number of participants with a discontinuation or temporary suspension of study drugs (for any reason) | 29 days
Cumulative incidence of AEs of Special Interest | 29 days

OTHER OUTCOMES:
Percent of subjects with SARS-CoV-2 detectable in nasopharyngeal sample | Days 3, 5, 8, 11, 15, 29
Quantitative SARS-CoV-2 virus in nasopharyngeal sample | Days 3, 5, 8, 11, 15, 29
Quantitative SARS-CoV-2 virus in blood | Days 3, 8

CONTACTS AND LOCATIONS:
Overall Officials: Florence Ader, MD, Study Chair — Hospices Civils de Lyon
Locations (60):
- Austria (3):
  - Medizinische Universität Innsbruck, Innsbruck
  - Kepler Universitätsklinikum Linz, Linz
  - Landeskrankenhaus Salzburg Universitätsklinikum der Paracelsus Medizinischen Privatuniversität, Salzburg
- Belgium (4):
  - Hôpital Erasme - Cliniques universitaires de Bruxelles, Brussels
  - Hôpital Saint Luc, Brussels
  - Hôpital La Citadelle, Liège
  - Pôle Hospitalier Jolimont / site de Mons-Warquignies, Mons
- France (43):
  - Centre Hospitalier Universitaire Amiens-Picardie, Amiens
  - Centre Hospitalier Regional Metz-Thionville, Ars-Laquenexy
  - Centre Hospitalier Régional Universitaire de Besançon, Besançon
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - CHU APHP Ambroise-Paré, Boulogne-Billancourt
  - Centre Hospitalier Andrée Rosemon, Cayenne
  - Hospices Civil, Colmar
  - APHP - hôpital Henri-Mondor, Créteil
  - Centre Hospitalier Universitaire Dijon-Bourgogne, Dijon
  - Centre Hospitalier Annecy Genevois, Épagny
  - Centre Hospitalier Universitaire de Martinique, Fort de France
  - Centre Hospitalo-Universitaire de Grenoble, La Tronche
  - AP-HP Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Groupe Hospitalier de la Région de Mulhouse Sud Alsace, Mulhouse
  - Centre Hospitalier Régional et Universitaire de Nancy, Nancy
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hospitalo-Universitaire de Nice, Nice
  - CHU Nîmes, Nîmes
  - APHP - Hôpital Lariboisière, Paris
  - APHP - Hôpital Saint Louis, Paris
  - APHP - Hôpital Saint Antoine, Paris
  - APHP - Hôpital Universitaire Pitié Salpêtrière, Paris
  - APHP - Hôpital Cochin, Paris
  - Hôpital Paris Saint-Joseph et Marie Lannelongue, Paris
  - APHP - Hôpital Necker, Paris
  - APHP- Hôpital Européen Georges-Pompidou, Paris
  - APHP - Hôpital Bichat Claude Bernard, Paris
  - APHP - Hôpital Tenon, Paris
  - CHU Poitiers, Poitiers
  - CH Cornouaille, Quimper
  - CHU de Reims, Reims
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Hopital DELAFONTAINE, Saint-Denis
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Etienne
  - Hôpital d'Instruction des Armées BEGIN, Saint-Mandé
  - Centre Hospitalier Régional Universitaire de Strasbourg, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
  - Centre Hospitalier de Tourcoing, Tourcoing
  - Centre Hospitalier Universitaire de Tours, Tours
  - CH Bretagne Atlantique, Vannes
- Greece (2):
  - Evaggelismos General Hospital, Athens
  - General University Hospital of Patras, Pátrai
- Luxembourg (2):
  - Centre Hospitalier Luxembourg, Luxembourg
  - Hôpitaux Robert Schuman, Luxembourg
- Norway (3):
  - Akershus Unniversity Hospital, Oslo
  - Lovisenberg Diaconal Hospital, Oslo
  - Oslo University Hospital, Oslo
- Portugal (3):
  - Hospital de Cascais, Cascais
  - CHULN- Hospital de Santa Maria, Lisbon
  - Centro Hospitalar Universitário de São João, EPE, Porto

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan will be available. Systematic individual patient data sharing is not intended, but all requests for the trial's data will be considered by the French DisCoVeRy Trial Management Team.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and statistical analysis plan will be available from September 2020 with no time limit.
  Other data will be available upon request after first publication of the results for at least 5 years
Access Criteria: Study protocol and statistical analysis plan will be published. All requests for the trial's data will be considered by the French DisCoVeRy Trial Management Team that can be contacted via the principal investigator: florence.ader@chu-lyon.fr

REFERENCES:
- [Background] Ader F; Discovery French Trial Management Team. Protocol for the DisCoVeRy trial: multicentre, adaptive, randomised trial of the safety and efficacy of treatments for COVID-19 in hospitalised adults. BMJ Open. 2020 Sep 21;10(9):e041437. doi: 10.1136/bmjopen-2020-041437. PMID 32958495
- [Background] EU-Response investigators group; Diallo A, Troseid M, Simensen VC, Boston A, Demotes J, Olsen IC, Chung F, Paiva JA, Hites M, Ader F, Arribas JR, Baratt-Due A, Melien O, Tacconelli E, Staub T, Greil R, Tsiodras S, Briel M, Esperou H, Mentre F, Eustace J, Saillard J, Delmas C, LeMestre S, Dumousseaux M, Costagliola D, Rottingen JA, Yazdanpanah Y. Accelerating clinical trial implementation in the context of the COVID-19 pandemic: challenges, lessons learned and recommendations from DisCoVeRy and the EU-SolidAct EU response group. Clin Microbiol Infect. 2022 Jan;28(1):1-5. doi: 10.1016/j.cmi.2021.10.011. Epub 2021 Nov 8. No abstract available. PMID 34763056
- [Background] Troseid M, Hentzien M, Ader F, Cardoso SW, Arribas JR, Molina JM, Mueller N, Hites M, Bonnet F, Manuel O, Costagliola D, Grinsztejn B, Olsen IC, Yazdapanah Y, Calmy A; EU RESPONSE; COMBINE. Immunocompromised patients have been neglected in COVID-19 trials: a call for action. Clin Microbiol Infect. 2022 Sep;28(9):1182-1183. doi: 10.1016/j.cmi.2022.05.005. Epub 2022 May 25. No abstract available. PMID 35623577
- [Background] Terzic V, Levoyer L, Figarella M, Bigagli E, Mercier N, De Gastines L, Gibowski S, Troseid M, Demotes J, Olsen IC, Hites M, Ader F, Lopez JRA, Mentre F, Esperou H, Costagliola D, Rottingen JA, Poissy J, Roze JC, Warris A, O'Leary J, Fernandes RM, Assoumou L, Hankard R, Turner MA, Yazdanpanah Y, Diallo A; EU-Response safety group; c4c safety group. Implementation of a centralized pharmacovigilance system in academic pan-European clinical trials: Experience from EU-Response and conect4children consortia. Br J Clin Pharmacol. 2023 Apr;89(4):1318-1328. doi: 10.1111/bcp.15669. Epub 2023 Feb 8. PMID 36680782
- [Background] Amstutz A, Speich B, Mentre F, Rueegg CS, Belhadi D, Assoumou L, Burdet C, Murthy S, Dodd LE, Wang Y, Tikkinen KAO, Ader F, Hites M, Bouscambert M, Trabaud MA, Fralick M, Lee TC, Pinto R, Barratt-Due A, Lund-Johansen F, Muller F, Nevalainen OPO, Cao B, Bonnett T, Griessbach A, Taji Heravi A, Schonenberger C, Janiaud P, Werlen L, Aghlmandi S, Schandelmaier S, Yazdanpanah Y, Costagliola D, Olsen IC, Briel M. Effects of remdesivir in patients hospitalised with COVID-19: a systematic review and individual patient data meta-analysis of randomised controlled trials. Lancet Respir Med. 2023 May;11(5):453-464. doi: 10.1016/S2213-2600(22)00528-8. Epub 2023 Feb 21. PMID 36828006
- [Background] Le MP, Peiffer-Smadja N, Guedj J, Neant N, Mentre F, Ader F, Yazdanpanah Y, Peytavin G. Rationale of a loading dose initiation for hydroxychloroquine treatment in COVID-19 infection in the DisCoVeRy trial. J Antimicrob Chemother. 2020 Sep 1;75(9):2376-2380. doi: 10.1093/jac/dkaa191. PMID 32473020
- [Background] Le MP, Peiffer-Smadja N, Guedj J, Neant N, Mentre F, Ader F, Yazdanpanah Y, Peytavin G; C-20-15 DisCoVeRy French Steering Committee. Rationale of a loading dose initiation for hydroxychloroquine treatment in COVID-19 infection in the DisCoVeRy trial-authors' response. J Antimicrob Chemother. 2021 Jan 1;76(1):277-279. doi: 10.1093/jac/dkaa415. No abstract available. PMID 33089306
- [Background] Mercier N, Belhadi D, DeChanet A, Delmas C, Saillard J, Dumousseaux M, Le Mestre S, Fougerou-Leurent C, Ferrane A, Burdet C, Esperou H, Ader F, Hites M, Peiffer-Smadja N, Poissy J, Andrejak C, Paiva JA, Tacconelli E, Staub T, Greil R, Costagliola D, Mentre F, Yazdanpanah Y, Diallo A; DisCoVeRy Safety Working group. Management of pharmacovigilance during the COVID-19 pandemic crisis by the safety department of an academic sponsor: Lessons learnt and challenges from the EU DisCoVeRy clinical trial. Pharmacol Res Perspect. 2023 Jun;11(3):e01072. doi: 10.1002/prp2.1072. PMID 37269068
- [Background] Fougerou-Leurent C, Delmas C, Saillard J, Dumousseaux M, Ferrane A, Mercier N, Terzic V, Le Mestre S, Dechanet A, Belhadi D, Metois A, Burdet C, Mentre F, Noret M, Diallo A, Petrov-Sanchez V, Couffin-Cadiergues S, Hites M, Ader F, Esperou H. Ensuring quality control in a COVID-19 clinical trial during the pandemic: The experience of the Inserm C20-15 DisCoVeRy study. Contemp Clin Trials. 2023 Aug;131:107267. doi: 10.1016/j.cct.2023.107267. Epub 2023 Jun 9. PMID 37302469
- [Background] Beaulieu M, Gaymard A, Massonnaud C, Peiffer-Smadja N, Bouscambert-Duchamp M, Carcelain G, Lingas G, Mentre F, Ader F, Hites M, Poignard P, Guedj J. Antiviral effect of Evusheld in COVID-19 hospitalized patients infected with pre-Omicron or Omicron variants: a modelling analysis of the randomized DisCoVeRy trial. J Antimicrob Chemother. 2024 Nov 4;79(11):2887-2895. doi: 10.1093/jac/dkae301. PMID 39236218
- [Background] Siempos II, Kalil AC, Belhadi D, Veiga VC, Cavalcanti AB, Branch-Elliman W, Papoutsi E, Gkirgkiris K, Xixi NA, Kotanidou A, Hermine O, Porcher R, Mariette X; CORIMUNO-19 Collaborative Group; DisCoVeRy Study Group; ACTT-2 Study Group; ACTT-3 Study Group. Immunomodulators for immunocompromised patients hospitalized for COVID-19: a meta-analysis of randomized controlled trials. EClinicalMedicine. 2024 Feb 9;69:102472. doi: 10.1016/j.eclinm.2024.102472. eCollection 2024 Mar. PMID 38361992
- [Result] WHO Solidarity Trial Consortium; Pan H, Peto R, Henao-Restrepo AM, Preziosi MP, Sathiyamoorthy V, Abdool Karim Q, Alejandria MM, Hernandez Garcia C, Kieny MP, Malekzadeh R, Murthy S, Reddy KS, Roses Periago M, Abi Hanna P, Ader F, Al-Bader AM, Alhasawi A, Allum E, Alotaibi A, Alvarez-Moreno CA, Appadoo S, Asiri A, Aukrust P, Barratt-Due A, Bellani S, Branca M, Cappel-Porter HBC, Cerrato N, Chow TS, Como N, Eustace J, Garcia PJ, Godbole S, Gotuzzo E, Griskevicius L, Hamra R, Hassan M, Hassany M, Hutton D, Irmansyah I, Jancoriene L, Kirwan J, Kumar S, Lennon P, Lopardo G, Lydon P, Magrini N, Maguire T, Manevska S, Manuel O, McGinty S, Medina MT, Mesa Rubio ML, Miranda-Montoya MC, Nel J, Nunes EP, Perola M, Portoles A, Rasmin MR, Raza A, Rees H, Reges PPS, Rogers CA, Salami K, Salvadori MI, Sinani N, Sterne JAC, Stevanovikj M, Tacconelli E, Tikkinen KAO, Trelle S, Zaid H, Rottingen JA, Swaminathan S. Repurposed Antiviral Drugs for Covid-19 - Interim WHO Solidarity Trial Results. N Engl J Med. 2021 Feb 11;384(6):497-511. doi: 10.1056/NEJMoa2023184. Epub 2020 Dec 2. PMID 33264556
- [Result] Ader F, Peiffer-Smadja N, Poissy J, Bouscambert-Duchamp M, Belhadi D, Diallo A, Delmas C, Saillard J, Dechanet A, Mercier N, Dupont A, Alfaiate T, Lescure FX, Raffi F, Goehringer F, Kimmoun A, Jaureguiberry S, Reignier J, Nseir S, Danion F, Clere-Jehl R, Bouiller K, Navellou JC, Tolsma V, Cabie A, Dubost C, Courjon J, Leroy S, Mootien J, Gaci R, Mourvillier B, Faure E, Pourcher V, Gallien S, Launay O, Lacombe K, Lanoix JP, Makinson A, Martin-Blondel G, Bouadma L, Botelho-Nevers E, Gagneux-Brunon A, Epaulard O, Piroth L, Wallet F, Richard JC, Reuter J, Staub T, Lina B, Noret M, Andrejak C, Le MP, Peytavin G, Hites M, Costagliola D, Yazdanpanah Y, Burdet C, Mentre F; DisCoVeRy study group. An open-label randomized controlled trial of the effect of lopinavir/ritonavir, lopinavir/ritonavir plus IFN-beta-1a and hydroxychloroquine in hospitalized patients with COVID-19. Clin Microbiol Infect. 2021 Dec;27(12):1826-1837. doi: 10.1016/j.cmi.2021.05.020. Epub 2021 May 26. PMID 34048876
- [Result] Ader F, Bouscambert-Duchamp M, Hites M, Peiffer-Smadja N, Poissy J, Belhadi D, Diallo A, Le MP, Peytavin G, Staub T, Greil R, Guedj J, Paiva JA, Costagliola D, Yazdanpanah Y, Burdet C, Mentre F; DisCoVeRy Study Group. Remdesivir plus standard of care versus standard of care alone for the treatment of patients admitted to hospital with COVID-19 (DisCoVeRy): a phase 3, randomised, controlled, open-label trial. Lancet Infect Dis. 2022 Feb;22(2):209-221. doi: 10.1016/S1473-3099(21)00485-0. Epub 2021 Sep 14. PMID 34534511
- [Result] Lingas G, Neant N, Gaymard A, Belhadi D, Peytavin G, Hites M, Staub T, Greil R, Paiva JA, Poissy J, Peiffer-Smadja N, Costagliola D, Yazdanpanah Y, Wallet F, Gagneux-Brunon A, Mentre F, Ader F, Burdet C, Guedj J, Bouscambert-Duchamp M. Effect of remdesivir on viral dynamics in COVID-19 hospitalized patients: a modelling analysis of the randomized, controlled, open-label DisCoVeRy trial. J Antimicrob Chemother. 2022 Apr 27;77(5):1404-1412. doi: 10.1093/jac/dkac048. PMID 35233617
- [Result] Ader F, Bouscambert-Duchamp M, Hites M, Peiffer-Smadja N, Mentre F, Burdet C; DisCoVeRy Study Group. Final results of the DisCoVeRy trial of remdesivir for patients admitted to hospital with COVID-19. Lancet Infect Dis. 2022 Jun;22(6):764-765. doi: 10.1016/S1473-3099(22)00295-X. No abstract available. PMID 35643099
- [Result] Ader F; DisCoVeRy Study Group. An open-label randomized, controlled trial of the effect of lopinavir and ritonavir, lopinavir and ritonavir plus interferon-beta-1a, and hydroxychloroquine in hospitalized patients with COVID-19: final results. Clin Microbiol Infect. 2022 Sep;28(9):1293-1296. doi: 10.1016/j.cmi.2022.04.016. Epub 2022 May 7. No abstract available. PMID 35533972
- [Result] Neant N, Lingas G, Gaymard A, Belhadi D, Hites M, Staub T, Greil R, Paiva JA, Poissy J, Peiffer-Smadja N, Costagliola D, Yazdanpanah Y, Bouscambert-Duchamp M, Gagneux-Brunon A, Ader F, Mentre F, Wallet F, Burdet C, Guedj J; DisCoVeRy study group. Association between SARS-CoV-2 viral kinetics and clinical score evolution in hospitalized patients. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2027-2037. doi: 10.1002/psp4.13051. Epub 2023 Oct 11. PMID 37728045
- [Result] WHO Solidarity Trial Consortium. Remdesivir and three other drugs for hospitalised patients with COVID-19: final results of the WHO Solidarity randomised trial and updated meta-analyses. Lancet. 2022 May 21;399(10339):1941-1953. doi: 10.1016/S0140-6736(22)00519-0. Epub 2022 May 2. PMID 35512728
- [Result] Hites M, Massonnaud CR, Lapique EL, Belhadi D, Jamard S, Goehringer F, Danion F, Reignier J, de Castro N, Garot D, Lacombe K, Tolsma V, Faure E, Malvy D, Staub T, Courjon J, Cazenave-Roblot F, Dyrhol Riise AM, Leturnier P, Martin-Blondel G, Roger C, Akinosoglou K, Moing VL, Piroth L, Sellier P, Lescure X, Troseid M, Clevenbergh P, Dalgard O, Gallien S, Gousseff M, Loubet P, Vardon-Bounes F, Visee C, Belkhir L, Botelho-Nevers E, Cabie A, Kotanidou A, Lanternier F, Rouveix-Nordon E, Silva S, Thiery G, Poignard P, Carcelain G, Diallo A, Mercier N, Terzic V, Bouscambert-Duchamp M, Gaymard A, Trabaud MA, Destras G, Josset L, Billard N, Han TH, Guedj J, Couffin-Cadiergues S, Dechanet A, Delmas C, Esperou H, Fougerou-Leurent C, Mestre SL, Metois A, Noret M, Bally I, Dergan-Dylon S, Tubiana S, Kalif O, Bergaud N, Leveau B, Eustace J, Greil R, Hajdu E, Halanova M, Paiva JA, Piekarska A, Rodriguez Bano J, Tonby K, Trojanek M, Tsiodras S, Unal S, Burdet C, Costagliola D, Yazdanpanah Y, Peiffer-Smadja N, Mentre F, Ader F; DisCoVeRy study group. Tixagevimab-cilgavimab (AZD7442) for the treatment of patients hospitalized with COVID-19 (DisCoVeRy): A phase 3, randomized, double-blind, placebo-controlled trial. J Infect. 2024 Mar;88(3):106120. doi: 10.1016/j.jinf.2024.106120. Epub 2024 Feb 16. No abstract available. PMID 38367705
- [Result] Terzic V, Miantezila Basilua J, Billard N, de Gastines L, Belhadi D, Fougerou-Leurent C, Peiffer-Smadja N, Mercier N, Delmas C, Ferrane A, Dechanet A, Poissy J, Esperou H, Ader F, Hites M, Andrejak C, Greil R, Paiva JA, Staub T, Tacconelli E, Burdet C, Costagliola D, Mentre F, Yazdanpanah Y, Diallo A; DisCoVeRy Study Group. Cardiac Adverse Events and Remdesivir in Hospitalized Patients With COVID-19: A Post Hoc Safety Analysis of the Randomized DisCoVeRy Trial. Clin Infect Dis. 2024 Aug 16;79(2):382-391. doi: 10.1093/cid/ciae170. PMID 38552208
- [Derived] Grundeis F, Ansems K, Dahms K, Thieme V, Metzendorf MI, Skoetz N, Benstoem C, Mikolajewska A, Griesel M, Fichtner F, Stegemann M. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2023 Jan 25;1(1):CD014962. doi: 10.1002/14651858.CD014962.pub2. PMID 36695483
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Ansems K, Grundeis F, Dahms K, Mikolajewska A, Thieme V, Piechotta V, Metzendorf MI, Stegemann M, Benstoem C, Fichtner F. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD014962. doi: 10.1002/14651858.CD014962. PMID 34350582
- [Derived] Taccone FS, Gorham J, Vincent JL. Hydroxychloroquine in the management of critically ill patients with COVID-19: the need for an evidence base. Lancet Respir Med. 2020 Jun;8(6):539-541. doi: 10.1016/S2213-2600(20)30172-7. Epub 2020 Apr 15. No abstract available. PMID 32304640